CLINICAL TRIAL: NCT01270334
Title: Effect of Vaginal PH on Treatment Effectiveness With Misoprostol for First Trimester Missed Abortions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: doctor baram shira, HaEmek Medical Center
Other Study IDs: cytoph
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2011-01

CONDITIONS: MISED ABORTION- Vaginal PH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ph above cutoff
  Interventions: Other: PH meassurment
- PH under cutoff
  Interventions: Other: PH meassurment

INTERVENTIONS:
Other: PH meassurment — meassuring ph USING PROBE

SUMMARY:
vaginal PH has an effect on the effectiveness of treatment with misoprostol given vaginally for missed abortions in the first trimester

ELIGIBILITY:
Inclusion

* missed abortion under 8 weeks by sac diameter over 18 years old informed concent given

Exclusion Criteria:

* missed abortion over 8 weeks hypersensitivity for PG vaginal bleeding suspected EUP IUD heart disease, HTN, cerebral vascular disease, epilepsy intrauterine infection clooting disorder under 18

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women dignosed with missed abortion in the first trimester
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-02

PRIMARY OUTCOMES:
treatment failure- need for D&C | 2 weeks

SECONDARY OUTCOMES:
side effects, need foe analgetics, time for compliting abortion | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Haemel Medical Center, Afula, Israel